CLINICAL TRIAL: NCT02394821
Title: Odor Management in Fungating Wounds Comparing Metronidazole and Polihexanide: Randomized Clinical Trial
Brief Title: Odor Management in Fungating Wounds Comparing Metronidazole and Polihexanide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, DIANA LIMA VILLELA DE CASTRO, ODOR MANAGEMENT IN FUNGATING WOUDS WITH METRONIDAZOLE versus PHMB: DOUBLE-BLINDED, RANDOMIZED, CLINICAL TRIAL, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: EE-USP5571275
Record Dates: First submitted 2014-05-08; First posted 2015-03-20 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Neoplasm; Wounds and Injuries
MeSH Terms: conditions — Neoplasms; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronidazole (Experimental): metronidazole 0.8% solution - topical
  Interventions: Drug: Metronidazole 0.8%
- Polihexanide (Experimental): Polihexanide 2%
  Interventions: Drug: Polihexanide 2%

INTERVENTIONS:
Drug: Polihexanide 2%
  Arms: Polihexanide
Drug: Metronidazole 0.8%
  Arms: Metronidazole

SUMMARY:
For odor control malignant wounds (MW), use is 0.8% metronidazole solution - second recommendation scientific and clinical practice. But no this formulation available in Brazil , and its application to nursing steeps metronidazole tablets , diluted in saline and applied to the bed of (MW) . Thus , it is used off label for metronidazole ( tablets orally applied via " topical " - but it is not intact skin or mucosa ) , nursing and eventually manipulate the solution at bedside , and by law this power is pharmacist bedside and can not be taken .

Family antiseptic chlorhexidine was developed with the purpose of use in infected wounds called polihexanide ( PHMB ) . In Brazil is now available for hospital and home care ( 0.2 % Aquasept ® ) use. Evidence reported positive results in controlling infection of chronic wounds such as pressure ulcers . Although not tested its efficacy in odor control. Thus the study aims to compare metronidazole solution 0.8 % versus 0.2 % PHMB in odor control , where , if the results are favorable to PHMB we have a treatment option in odor control with ready to use formulation and easy access . Evaluate and compare the effectiveness of metronidazole solution 0.8% and polihexanide solution (PHMB) in odor control in MW. Aims: Evaluate and compare the time needed for odor control (reduction in days), using metronidazole and PHMB in MW (primary endpoint); Evaluate and compare the perceptions of patients, nurses and researcher on the odor MW, using metronidazole and PHMB in the MW; Evaluate and compare the pain reported by patients during dressing changes, using metronidazole and PHMB in the MW; Evaluate and compare the quality of life of patients before and after the use of metronidazole and PHMB in MW. This is a randomized, double -blind study with patients diagnosed with cancer and patients with MW with odor clinical trial . The sample consisted of 24 subjects divided into 2 groups (control - metronidazole group and experimental group - PHMB ) , recruited in one cancer hospital in the city of São Paulo (AC Camargo Cancer Center), which has as protocol description in odor control MW metronidazole . After acceptance by the subject and return the Statement of Informed Consent signed , randomization will be done .

For blinding , 0.8 % metronidazole solution will be provided by a compounding pharmacy (after stability testing of tablet diluted - and then stipulated expiration date) , and PHMB be bought from the supplier , delivered to the same compounding pharmacy which stores the PHMB in identical bottles to metronidazole ( only the responsible researcher will know to which group the subject was randomized ) .

The evaluation of the odor will be taken by 3 " employees " and the patient through 3 scales at zero , four, eight and twelve days ( or earlier if classified as " odorless " by 3 reviewers and the patient ) . Two scales about painful sensations in exchange for healing , one on quality of life will be applied to the patient and a specifically on the impact of odor on the subject's life.

To meet the proposed objectives, the data will be analyzed by: Friedman test to assess the odor reduction with respect to time; Mann-Whitney (or t test) for comparison of groups and the Fisher exact test to compare proportions. Data will be presented in the form of frequency tables for categorical variables and means, standard deviations and position measurements for quantitative variables. Will also be performed non-parametric analysis of ordinal data, or parametric analysis with Generalized Estimation Equation for binomial variables, depending on the data distribution and the sample size.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of malignat wound with odor, regardless of location, etiology and tumor staging; well as in treatment or palliative care.
* Confirmation of participation in the study by signing the Instrument of Consent, personally or through responsible caretaker

Exclusion Criteria:

* not smell

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Evaluate and compare the effectiveness of metronidazole solution 0.8% and polihexanide solution (PHMB) in odor control in malignant wounds. (odor scales) | 30/12/2014 (up to 1 year)

SECONDARY OUTCOMES:
To evaluate and compare the time required for odor control (reductions in days), using metronidazole and PHMB in malignant wounds (Friedman test to assess the odor reduction with respect to time) | 30/12/2014 (up to 1 year)

OTHER OUTCOMES:
Evaluate and compare the perceptions of patients, nurses and researcher on the odor in malignant wounds, using metronidazole and PHMB in malignant wounds; (evaluation of odor scales [painful sensations in exchange for healing , and quality of life]) | 30/12/2014 (up to 1 year)

CONTACTS AND LOCATIONS:
Locations (1):
- EEUSP, São Paulo, São Paulo, Brazil